CLINICAL TRIAL: NCT04063306
Title: Investigation on Quality of Life and Related Factors of Taiwan People Living With HIV
Brief Title: Quality of Life of Taiwan People Living With HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taiwan AIDS Nurse Society (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Chung-Ching Shih, Research & Development Board Director, Taiwan AIDS Nurse Society
Other Study IDs: TANA-2019-01
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: none of intervention was given — this is an observational survey and no intervention is given

SUMMARY:
To survey QoL and relevant factors in PLWH

ELIGIBILITY:
Inclusion Criteria:

* adult patient living with HIV, aged >= 18 years old

Exclusion Criteria:

* known cognitive dysfunction or attention deficient to complete the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult HIV-1 infected patients
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-10-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
QoL status of Patient Living with HIV (PLWH) by WHOQOL-HIV Brief questionaire | in 4 weeks
Medical Outcome of Patient Living with HIV (PLWH) by MOS-HIV questionaire | in 4 weeks
Stigma Scale of Patient Living with HIV (PLWH) by Berger's HIV Stigma Scale | an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided